CLINICAL TRIAL: NCT02609672
Title: Resilience and Longevity for Older Workers With Arthritis Through Exercise
Brief Title: Resilience for Older Workers With OA Through Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ResilienceAtWork
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2017-09

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
Keywords: Exercise; Resilience
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (Experimental): The participants in this arm were asked to attend 3 group classes per week for 12 weeks taught by a certified exercise instructor. Four class times were offered per week. These classes included a warm-up, static poses shown to decrease knee joint loading, and a cool down including flexibility exercises. Measurements were obtained at baseline (before intervention) and at follow-up (following intervention). Outcomes included clinical mobility; pain; isometric leg strength; cardiovascular fitness; and resilience.
  Interventions: Other: Exercise
- No Exercise (Other): The participants in this arm were asked to refrain from changing their physical activity over the 12 weeks and maintain any strategies typically used to manage knee and/or hip pain. Since it is known that exercise is beneficial for pain management and strengthening in knee OA, participants randomized to the no exercise group were offered a free exercise pass following completion of the study. Measurements were obtained at baseline (before intervention) and at follow-up (following intervention). Outcomes included clinical mobility; pain; isometric leg strength; cardiovascular fitness; and resilience.
  Interventions: Other: No Exercise

INTERVENTIONS:
Other: Exercise — A biomechanical exercise program shown to decrease joint loading was administered 3 times a week for 12 weeks. Outcomes included mobility performance; pain; strength; cardiovascular fitness; and resilience.
  Arms: Exercise
Other: No Exercise — A no exercise (control) group maintained their existing activity level for 12 weeks. Outcomes included mobility performance; pain; strength; cardiovascular fitness; and resilience.
  Arms: No Exercise

SUMMARY:
Exercise is effective at reducing pain while improving physical function. However we do not know if exercise can boost resilience in the workplace, to allow people with osteoarthritis to work as long as they desire. Previous research shows that exercise holds the most promise for helping people enjoy their work because it reduces sick time, reduces pain, and improves productivity. However, little work has examined the effect of exercise for people with arthritis in the workplace. The purpose of the study is to investigate whether exercise improves resilience in the workplace, mobility, fitness, strength, and pain in comparison to no exercise in those with knee and/or hip osteoarthritis.

DETAILED DESCRIPTION:
The Canadian workforce is aging. The most prevalent age group is 50-54 years and most of these Canadians will aim to continue working over the next 10 years. However, the impact of arthritis on aging Canadians compromises their ability to continue working. By 2031, over 2 million Canadians aged 45 to 64 years will have arthritis. We aim to boost the ability of older adults with the most common arthritis, osteoarthritis (OA), to engage in the workforce for as long as they desire. Identifying strategies to promote productivity among older workers with knee and hip OA will be of great public health significance in the coming decades. However, we face two challenges. First, obesity among sedentary workers is a risk for worsening knee and hip OA. Second, large occupational loads on the knee and hip worsen OA. Exercise has the most promise in addressing these challenges because it reduces pain and sick time, and improves mental health. Thus, there is a call for studies examining exercise for the aging worker with knee and hip OA. The purpose of this study is to examine the impact of an OA-specific leg strengthening exercise program, delivered within the workplace, on mobility, pain, physical capacity, and resilience among older workers with knee or hip OA.

ELIGIBILITY:
Inclusion Criteria:

* 45 years of age or older
* McMaster employee
* Sedentary job (stand or walk for <1/3 of work day)
* Able to safely climb two flights of stairs
* Hip pain
* Hip pain during internal rotation and hip flexion
* Knee pain
* Less than 30 minutes of morning stiffness in the knee
* Crepitus in the knee with active range of motion
* Bony enlargement around the knee
* Bony tenderness to palpation at the knee
* No warmth around the knee

Exclusion Criteria:

* Any other forms of arthritis
* Osteoporosis-related fracture
* History of patellofemoral symptoms
* Active non-arthritic hip or knee disease
* Hip or knee surgery
* Use of cane or walking aid
* Unstable heart condition
* Neurological conditions
* Hip, knee or ankle injuries in past 3 months
* Physician-advised restriction to physical activity
* Any injuries that would prohibit participation in exercise
* Ipsilateral ankle conditions
* Currently receiving cancer treatment
* Currently pregnant

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica R Maly, PT, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chopp-Hurley JN, Brenneman EC, Wiebenga EG, Bulbrook B, Keir PJ, Maly MR. Randomized Controlled Trial Investigating the Role of Exercise in the Workplace to Improve Work Ability, Performance, and Patient-Reported Symptoms Among Older Workers With Osteoarthritis. J Occup Environ Med. 2017 Jun;59(6):550-556. doi: 10.1097/JOM.0000000000001020. PMID 28379878

RESULTS

PARTICIPANT FLOW:
Groups:
- No Exercise: The participants in this arm were asked to refrain from changing their physical activity over the 12 weeks and maintain any strategies typically used to manage knee and/or hip pain. Since it is known that exercise is beneficial for pain management and strengthening in knee osteoarthritis, participants randomized to the no exercise group were offered a free exercise pass following completion of the study. Measurements were obtained at baseline (before intervention) and at follow-up (following intervention). Outcomes included clinical mobility; pain; isometric leg strength; cardiovascular fitness; and resilience.
  No Exercise: A no exercise (control) group maintained their existing activity level for 12 weeks. Outcomes included mobility performance; pain; strength; cardiovascular fitness; and resilience.
Period: Overall Study
Arm/Group | Exercise | No Exercise
Started | 12 | 12
Completed | 9 | 11
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise | No Exercise | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (6.4) | 54.9 (6.7) | 53.9 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  Canada | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Lower Extremity Function
Description: The Lower Extremity Function Scale (LEFS) consists of 20 items, on an adjectival scale, that assess difficulty during mobility tasks ranging from transfers to running. Each item is scored from 0 (extreme difficulty or unable to perform activity), to 4 (no difficulty to perform activity). The minimum possible score is 0, and the maximum possible score is 80. Scores closer to 80 represent better self-reported physical function. It is reliable and valid in knee OA and has superior sensitivity to change compared to similar measures.
Time Frame: Week 1 and Week 13
Measure: Mean (Standard Deviation); unit: Change in scores on a scale
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 9 | 11
Change in scores on a scale | 6.9 (12.9) | 0.5 (10.6)

2. Secondary Outcome: Change in Self-reported Knee and Hip Pain
Description: Change in self-reported knee and hip pain will be assessed with 3 valid and reliable questionnaires: the Knee injury and Osteoarthritis Outcome Score (KOOS), the Hip disability and Osteoarthritis Outcome Score (HOOS), and the Intermittent and Constant Osteoarthritis Pain (ICOAP) score. The KOOS and HOOS pain scores represent a normalized score from 0 (extreme symptoms) to 100 (no symptoms). KOOS and HOOS scores closer to 100 indicate fewer symptoms. The ICOAP consists of two sub-scales: constant pain (5 items) and intermittent pain (6 items). The score from each subscale represents a normalized score from 0 (no pain) to 100 (extreme pain). ICOAP scores closer to 0 indicate less pain. The items from each subscale are averaged to produce a normalized ICOAP total score, ranging from 0 (no pain) to 100 (extreme pain).
Time Frame: Week 1 and Week 13
Measure: Mean (Standard Deviation); unit: Change in scores on a scale
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 9 | 11
Change in scores on a scale
  KOOS Pain | 8.3 (13.3) | -1.0 (6.4)
  HOOS Pain | 4.1 (7.3) | 0.2 (13.3)
  ICOAP Constant | -20.6 (23.1) | -2.3 (11.7)
  ICOAP Intermittent | -26.4 (17.2) | 3.3 (22.0)
  ICOAP Total Score | -23.8 (18.5) | 0.8 (15.0)

3. Secondary Outcome: Change in Resilience
Description: Resilience will be measured using the Resilience Scale 25 Survey, which is a 25-item questionnaire designed to evaluate a participants ability to adapt to stress and adversity. The test is scored out of 175 (scores ranging from 25 to 175), with higher scores indicating higher resilience.
Time Frame: Week 1 and Week 13
Measure: Mean (Standard Deviation); unit: Change in scores on a scale
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 9 | 11
Change in scores on a scale | 6.2 (16.5) | 2.8 (10.4)

4. Secondary Outcome: Change in Mobility Performance (Six-Minute Walk Test)
Description: Mobility performance will be measured using the Six-Minute Walk Test (6MWT). For this test, participants are instructed to walk as far as possible in 6 minutes. The distance covered in 6 minutes is recorded in metres. This measure has produced reliable and valid data in persons with knee OA.
Time Frame: Week 1 and Week 13
Measure: Mean (Standard Deviation); unit: Change in Metres
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 9 | 11
Change in Metres | 12.5 (39.6) | 23.7 (54.1)

5. Secondary Outcome: Change in Mobility Performance (40 Metre Walk Test)
Description: Mobility performance will be measured using the 40 Metre Walk Test. This test measures the time taken to complete a fast-paced 40 metre walk. The time taken to walk 40 metres is recorded in seconds. This measure has produced reliable and valid data in persons with knee OA.
Time Frame: Week 1 and Week 13
Measure: Mean (Standard Deviation); unit: Change in Seconds
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 9 | 11
Change in Seconds | -0.7 (2.7) | -0.1 (2.4)

6. Secondary Outcome: Change in Mobility Performance (Stair Ascent)
Description: Mobility performance will be measured using the Stair Ascent Test. For this test, the time taken to ascend nine stairs is recorded in seconds. This measure has produced reliable and valid data in persons with knee OA.
Time Frame: Week 1 and Week 13
Measure: Mean (Standard Deviation); unit: Change in Seconds
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 9 | 11
Change in Seconds | -0.4 (0.6) | 0.0 (0.6)

7. Secondary Outcome: Change in Mobility Performance (Stair Descent)
Description: Mobility performance will be measured using the Stair Descent Test. For this test, the time taken to descend nine stairs is recorded in seconds. This measure has produced reliable and valid data in persons with knee OA.
Time Frame: Week 1 and Week 13
Measure: Mean (Standard Deviation); unit: Change in Seconds
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 9 | 11
Change in Seconds | -0.1 (0.4) | 0.0 (0.6)

8. Secondary Outcome: Change in Mobility Performance (30-second Chair Stand Test)
Description: Mobility performance will be measured using the 30-second Chair Stand Test. This test measures the number of times participants can rise and lower from a standard height chair, without using arm rests, in a 30-second period.This measure has produced reliable and valid data in persons with knee OA.
Time Frame: Week 1 and Week 13
Measure: Mean (Standard Deviation); unit: Change in number of sit-to-stand cycles
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 9 | 11
Change in number of sit-to-stand cycles | 0.2 (2.4) | -0.5 (2.5)

9. Secondary Outcome: Change in Mobility Performance (Timed Up and Go Test)
Description: Mobility performance will be measured using the Timed Up and Go Test. This test measures the time taken to rise from a standard chair with arm rests, walk 3 metres, and return to a seated position. This measure has produced reliable and valid data in persons with knee OA.
Time Frame: Week 1 and Week 13
Measure: Mean (Standard Deviation); unit: Change in Seconds
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 9 | 11
Change in Seconds | -0.5 (1.0) | 0.2 (1.0)

10. Secondary Outcome: Change in Arthritis-related Self-efficacy
Description: The Arthritis Self-Efficacy Scale (ASES) measures arthritis-specific beliefs regarding perception of performance on certain tasks to cope with the disease. The ASES is measured using 20 questions on a 10-100 scale with respect to three main areas: pain management (5 questions), physical function (9 questions), and other symptoms (6 questions). Each question is scored from 10 (very uncertain), to 100 (very certain), in 10-point increments. The minimum score for each subscale is 10, and the maximum score for each subscale is 100. The scores from each subscale are averaged to produce a normalized total score. Scores closer to 100 indicate greater certainty that a participant can cope with a particular task as a consequence of their disease.
Time Frame: Week 1 and Week 13
Measure: Mean (Standard Deviation); unit: Change in scores on a scale
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 9 | 11
Change in scores on a scale
  ASES Pain | 1.1 (2.5) | 0.6 (2.0)
  ASES Function | 0.9 (1.4) | 0.1 (0.7)
  ASES Symptoms | 1.6 (2.2) | 0.9 (1.5)
  ASES Total | 3.7 (5.6) | 1.6 (3.2)

11. Secondary Outcome: Change in Depression Status
Description: Depression will be assessed with the Centre of Epidemiological Studies Depression (CES-D) Scale, a 20-item scale developed for the general population with emphasis on affect. Elements of affect include mood, guilt, worthlessness, helplessness, appetite, and sleep. Each item is scored from 0 (rarely or none of the time), to 3 (most of the time). The items are summed to produce a total score between 0 and 60 with a score of 16 or higher indicating depression.
Time Frame: Week 1 and Week 13
Measure: Mean (Standard Deviation); unit: Change in scores on a scale
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 9 | 11
Change in scores on a scale | -7.2 (8.0) | 0.3 (6.1)

12. Secondary Outcome: Change in Grip Strength (Absolute)
Description: Grip strength will be assessed using a Jamar hand dynamometer. The hand dynamometer will be set to a fixed position and all values of grip force will be expressed in kg.
Time Frame: Week 1 and Week 13
Measure: Mean (Standard Deviation); unit: Change in kg
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 9 | 11
Change in kg
  Right Side Grip Strength | 1.1 (2.6) | -0.1 (2.8)
  Left Side Grip Strength | 0.4 (3.0) | -0.2 (2.8)

13. Secondary Outcome: Change in Grip Strength (Relative)
Description: Grip strength will be assessed using a Jamar hand dynamometer. The hand dynamometer will be set to a fixed position and all values of grip force will be expressed in kg/kg (grip force/body mass).
Time Frame: Week 1 and Week 13
Measure: Mean (Standard Deviation); unit: Change in kg/kg
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 9 | 11
Change in kg/kg
  Right Side Normalized Grip Strength | 0.0 (0.0) | 0.0 (0.0)
  Left Side Normalized Grip Strength | 0.0 (0.0) | 0.0 (0.0)

14. Secondary Outcome: Change in Isometric Knee and Hip Extensor and Flexor Strength
Description: The peak torque developed during knee and hip extension and flexion during a maximum isometric contraction will be measured by use of a Biodex System 2 isokinetic dynamometer. Data will be presented as Nm/kg (torque/body mass).
Time Frame: Week 1 and Week 13
Measure: Mean (Standard Deviation); unit: Change in Nm/kg
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 9 | 11
Change in Nm/kg
  Knee Extensor Torque (Nm/kg) | 0.1 (0.2) | -0.1 (0.2)
  Knee Flexor Torque (Nm/kg) | 0.0 (0.1) | 0.0 (0.1)
  Hip Extensor Torque (Nm/kg) | 0.1 (0.2) | 0.1 (0.2)
  Hip Flexor Torque (Nm/kg) | 0.0 (0.1) | 0.0 (0.1)

15. Secondary Outcome: Change in Cardiovascular Fitness
Description: Cardiovascular fitness will be calculated using the Single Stage Treadmill Walking Test. Predictions of VO2max will be made from heart rate (measured with a heart rate monitor), walking speed, age and gender.
Time Frame: Week 1 and Week 13
Population: Due to equipment problems, 2 participants from the Exercise Group were not able to complete the Single Stage Treadmill Walking Test.
Measure: Mean (Standard Deviation); unit: Change in ml/kg/min
Arm/Group | Exercise | No Exercise
Number analyzed (Participants) | 7 | 11
Change in ml/kg/min | -1.3 (3.0) | -1.7 (2.5)

ADVERSE EVENTS:
Arm/Group | Exercise | No Exercise
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
* Sample size in this trial was limited
* Adherence to the exercise classes in the exercise group was poor

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No